CLINICAL TRIAL: NCT06173154
Title: Feasibility Assessment of Implementing a Care System to PREVENT Iatrogenic Dependency (ID) Related to Hospitalization in People Over 70 Years : Pilot Study. PREVENT-ID
Brief Title: Feasibility Assessment of Implementing a Care System to PREVENT Iatrogenic Dependency (ID)
Acronym: PREVENT-ID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/21/0171
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Aged
Keywords: prevention; elderly; dependance; hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ID prevention unit (Experimental): One healthcare unit will implement the healthcare system for the prevention of iatrogenic dependency (ID) and one healthcare unit will provide standard care without any specific system in place.
  Interventions: Other: Care system to prevent ID
- Control unit (Sham Comparator): One healthcare unit will implement the healthcare system for the prevention of iatrogenic dependency (ID) and one healthcare unit will provide standard care without any specific system in place.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Care system to prevent ID — The caregivers of this unit receive training about iatrogenic dependency and how prevent it. They set up this prevention and the research compare evolution of dependence hospitalized patients.
  Arms: ID prevention unit
Other: Routine care — standard care without any specific system in place
  Arms: Control unit

SUMMARY:
To assess the feasibility of a care system to prevent iatrogenic dependency during hospitalisation in people 70 years old and over. 2 cares units participate : one with routine care and the other with a care system to prevent ID. The caregivers of this unit receive training about iatrogenic dependency and how prevent it. They set up this prevention and the research compare evolution of dependence hospitalized patients.

ELIGIBILITY:
inclusion criteria:

* Patient hospitalized for at least 48 hours in the participating center
* Persons affiliated to a social security system,
* The patient, his trusted person or a relative present during his hospitalization have not expressed opposition to his participation in the research..

exclusion criteria:

* End of life situation,
* ADL at 0/6 for 15 days before hospitalization.
* Refusal to participate,
* Patient under judicial protection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
number of participants with loss of independence | 15 days
  loss of independence is defined as a decrease of at least 0.5 points in Activities of Daily Living (ADL) scale between admission and discharge of the patient within 15 days of admission to the ward, regardless of when this event occurs during the hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline BERBON, Study Director — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No